CLINICAL TRIAL: NCT00881439
Title: A Double-blind, Placebo-controlled, Randomized Trial Investigating the Safety and Efficacy of Additive Renin Inhibition With Aliskiren on Renal Blood Flow and Neurohormonal Activation in Patients With Chronic Heart Failure and Renal Dysfunction
Brief Title: Safety and Efficacy Study of Add On Aliskiren in Patients With Heart Failure and Renal Impairment
Acronym: ARIANA-CHF-RD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, H.L. Hillege, Prof.dr., University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARIANA
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Heart Failure; Kidney Failure
Keywords: Heart failure; Renal Failure; Cardiorenal Syndrome; Renin inhibition; Aliskiren
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Cardio-Renal Syndrome | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Aliskiren (Active Comparator)
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — Oral, 300 mg, once daily, 6 months
  Other Names: Rasilez; SPP100
  Arms: Aliskiren
Drug: Placebo — Matching Placebo once daily, 6 months
  Arms: Placebo

SUMMARY:
The main purpose of this study is to examine the effect of add-on therapy with the direct renin inhibitor Aliskiren in comparison to placebo on renal blood flow in patients with heart failure and reduced renal function.

* Primary outcome measure: change in renal blood flow at 6 months
* Secondary outcome measures: changes in renal function, N-terminal pro Brain natriuretic peptide, left ventricular function, blood pressure and neurohormones

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo controlled, parallel group comparison trial, enrolling 100 patients (67 vs. 33) with stable CHF. Patients will be randomized to Aliskiren 300 mg once daily or corresponding Placebo for a period of 6 months. Efficacy measures will be performed at baseline and at the end of the study. Primary efficacy outcome is change in renal blood flow as measured by 131I-Hippuran clearance. Secondary outcome include change in renal function, neurohormones, left ventricular function and blood pressure. Safety assessments include renal function, changes in electrolytes, and blood pressure. Patients will be uptitrated to maximum tolerated doses of Aliskiren, and safety visits are planned 1 week after initiation and on a 2 month interval afterwards. A total of 8 visits are planned during the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* NYHA II-IV Heart Failure
* Left ventricular ejection fraction < 45%
* Stable heart failure medication
* eGFR by sMDRD formula between 30 and 60 mL/min/1.73m2

Exclusion Criteria:

* Known hypersensitivity to study drug or ACEi
* Concomitant treatment with both ARB and Aldosterone Receptor Antagonist
* Symptomatic Hypotension
* Acute Heart Failure
* History of stroke, acute coronary syndrome, PCI or angioplasty within past 3 months
* Serum potassium > 5.2 mmol/L
* Right heart failure due to severe pulmonary disease
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-04; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in renal blood flow as assessed by 131I-Hippuran clearance | 6 months

SECONDARY OUTCOMES:
change in glomerular filtration rate (GFR) as assessed by 125I-Iothalamate | 6 months
Change in systolic and diastolic blood pressure | 6 months
change in N-terminal pro brain natriuretic peptide levels (NT-proBNP) | 6 months
Change in left ventricular ejection fraction | 6 months
change in NYHA class, change in filtration fraction, change in albumin excretion, change in tubular function parameters, change in neurohormonal activation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] McMurray JJ, Pitt B, Latini R, Maggioni AP, Solomon SD, Keefe DL, Ford J, Verma A, Lewsey J; Aliskiren Observation of Heart Failure Treatment (ALOFT) Investigators. Effects of the oral direct renin inhibitor aliskiren in patients with symptomatic heart failure. Circ Heart Fail. 2008 May;1(1):17-24. doi: 10.1161/CIRCHEARTFAILURE.107.740704. PMID 19808266
- [Derived] Schroten NF, Damman K, Hemmelder MH, Voors AA, Navis G, Gaillard CA, van Veldhuisen DJ, Van Gilst WH, Hillege HL. Effect of additive renin inhibition with aliskiren on renal blood flow in patients with Chronic Heart Failure and Renal Dysfunction (Additive Renin Inhibition with Aliskiren on renal blood flow and Neurohormonal Activation in patients with Chronic Heart Failure and Renal Dysfunction). Am Heart J. 2015 May;169(5):693-701.e3. doi: 10.1016/j.ahj.2014.12.016. Epub 2015 Jan 7. PMID 25965717